CLINICAL TRIAL: NCT00004293
Title: Phase II Study of Glucocerebrosidase in Patients With Gaucher Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Pittsburgh (Other)
Purpose: Treatment
Other Study IDs: 199/11725; UPITTS-M1230
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Gaucher's Disease
Keywords: Gaucher's disease; inborn errors of metabolism; rare disease; sphingolipidoses
MeSH Terms: conditions — Gaucher Disease; Metabolism, Inborn Errors; Rare Diseases; Sphingolipidoses | interventions — Glucosylceramidase

INTERVENTIONS:
Drug: glucocerebrosidase

SUMMARY:
OBJECTIVES:

I. Evaluate the efficacy and toxicity of glucocerebrosidase enzyme therapy in patients with Gaucher disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are treated with intravenous glucocerebrosidase every 2 weeks. The dose is based on clinical severity of disease and response to therapy.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Gaucher disease with glucocerebrosidase deficiency confirmed by enzymatic or molecular assay At least 3 organ systems affected, based on the following criteria: Anemia Thrombocytopenia Organomegaly Bone deterioration on radiograph Pulmonary compromise Symptoms compromise daily activities or risk longevity No neurologic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: John Barranger, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States